CLINICAL TRIAL: NCT05090098
Title: Comparison of the Effects of Fear of Movement and Physical Activity Barriers on Physical Activity, Quality of Life and Psychological State of Women Who Have Had or Are Having Breast Cancer With Healthy People - Case Control Study
Brief Title: Breast Cancer and Kinesiophobia and Physical Activity
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Other Study IDs: ATADEK-2021/14/16
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Kinesiophobia
MeSH Terms: conditions — Breast Neoplasms; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer: Sixty patients with grade I-II-III breast cancer, whose primary treatment (surgery, radiotherapy and/or chemotherapy) is continuing, who applied to the Hospital Breast Unit clinic, will be included in the study. Patients with problems in reading and writing in Turkish, poor cognitive functions and a serious chronic disease, musculoskeletal pain or disease, severe psychiatric illness, current cancer attack or metastasis will be excluded from the study
  Interventions: Other: None intervention
- Breast cancer survivors: Sixty patients with grade I-II-III breast cancer, whose primary treatment (surgery, radiotherapy and/or chemotherapy) was completed at least three months ago, who applied to the Hospital Breast Unit clinic, will be included in the study. Patients with problems in reading and writing in Turkish, poor cognitive functions and a serious chronic disease, musculoskeletal pain or disease, severe psychiatric illness, current cancer attack or metastasis will be excluded from the study
  Interventions: Other: None intervention
- Healthy people: healthy individuals matched for age and gender will also be included in the study.
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention — None intervention

SUMMARY:
Breast cancer is the most common type of cancer in women worldwide. A significant number of breast cancer survivors develop many complications. Breast cancer and survivors may develop a fear of physical activity avoidance and movement, called kinesiophobia, due to upper extremity pain, numbness, restricted arm/shoulder range of motion, and risk of lymphedema. Therefore, in the present study, it is aimed to compare the effect of fear of movement on physical activity, quality of life and psychological states in women who have had breast cancer with healthy people.

ELIGIBILITY:
Inclusion Criteria:

* • Women diagnosed with stage I-II-III breast cancer with surgery as the first treatment

  * The patient whose first treatment was completed at least three months ago (surgery, radiotherapy and / or chemotherapy)
  * 18-75 years old woman
  * Does not have a Turkish literacy problem

Exclusion Criteria:

* • A serious chronic disease (rheumatoid arthritis, multiple sclerosis, amyotrophic lateral sclerosis, kidney disease, heart failure, neurological disorders or diabetes mellitus type I or II patients)

  * Having severe musculoskeletal pain or disease
  * Serious psychiatric illness
  * Patients with current cancer attack or metastasis
  * Persons with cognitive impairment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty patients with grade I-II-III breast cancer, whose primary treatment (surgery, radiotherapy and/or chemotherapy) was completed at least three months ago, who applied to the Acıbadem Maslak Hospital Breast Unit clinic, will be included in the study. Patients with problems in reading and writing in Turkish, poor cognitive functions and a serious chronic disease, musculoskeletal pain or disease, severe psychiatric illness, current cancer attack or metastasis will be excluded from the study [17]. Since it is a case-control study, 60 healthy individuals matched for age and gender will also be included in the study.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | Six month
  The TAMPA Kinesiophobia Scale consists of 17 questions. Each question is scored between 1-4. The maximum score is 68, with high scores indicating an increased severity of kinesiophobia. A score of more than 37 indicates high severity of kinesiophobia.
Questionnaire on exercise barriers | Six month
  This questionnaire contains a total of 35 obstacles. These obstacles are; symptom-related (n = 10), individual (n = 10), psychosocial (n = 8) and environmental (n = 7) factors. You will be asked if these obstacles prevent you from exercising.
INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRES (IPAQ) | Six month
  Physical activity level measured in Metabolic Equivalent

SECONDARY OUTCOMES:
Fatigue Severity Scale | Six month
  This scale consists of nine items. Each item is scored between 1 and 7, and as the total score decreases, fatigue decreases.
Hospital Anxiety and Depression Scale | Six month
  The lowest score that patients can get from both subscales is 0, and the highest score is 21. A high score indicates high anxiety and depression values.
Evaluation of Quality of Life: EORTC-Quality of Life -C 30 | Six month
  High scores indicate a high quality of life, and low scores indicate a decreased quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided